CLINICAL TRIAL: NCT03055052
Title: Clinical Effects of a Formula With Modified Protein Levels and Fat Blend in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 14.25.INF
Record Dates: First submitted 2017-01-26; First posted 2017-02-16 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Infant, Premature, Nutrition
MeSH Terms: conditions — Premature Birth | interventions — Food, Formulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Formula (Active Comparator): Standard formula for preterm infants.
  Interventions: Other: Standard formula for preterm infants
- Experimental formula (Experimental): Formula with higher protein and new fat blend for preterm infants.
  Interventions: Other: Formula with higher protein and new fat blend for preterm infants

INTERVENTIONS:
Other: Standard formula for preterm infants — Reconstituted in water and given to infants at more than 50% of feedings.
  Arms: Control Formula
Other: Formula with higher protein and new fat blend for preterm infants — Reconstituted in water and given to infants at more than 50% of feedings.
  Arms: Experimental formula

SUMMARY:
This study evaluates the effects of infant formula with higher protein level and improved fat blend on growth and feeding tolerance in preterm infants. Half of the subjects will receive a standard infant formula, while the other half will receive a infant formula with a higher protein level and improved fat blend.

DETAILED DESCRIPTION:
When an infant is born prematurely, the supply of nutrients supporting normal growth and development is interrupted. There is less time to accrue adequate nutrient stores and foetal tissue. The nutritional goal for the preterm infant is to have satisfactory functional development and catch up on growth to match the rate of a full term infant. To achieve this, it is recommended for the infant to have adequate protein intake and suitable fat blend.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 33 weeks 0 days
* Birth weight less than or equal to 2000g.
* Infant is anticipated to receive the study formula for ≥ 3 consecutive weeks
* At entry into Full Enteral Feeding, study formula will be provided at 50% or more of total enteral feedings.
* Written informed consent has been obtained from the parent/legally authorized representative (LAR).

Exclusion Criteria:

* Peri-/intra-ventricular hemorrhage
* Renal disease
* Hepatic dysfunction
* Major congenital malformations
* Suspected or documented systemic or congenital infections
* Cardiac, respiratory, endocrinologic, hematologic, GI, or other systemic diseases that may impact growth
* Suspected or documented maternal substance abuse
* Infants who have received any experimental treatment or intervention

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03-18 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Growth in terms of weight gain per day | 21 days

SECONDARY OUTCOMES:
Growth in terms of length and head circumference | Till infant reaches 3kg (study completion), expected within 3 months
Feeding tolerance (frequency of regurgitation, stool frequency and consistency) | Till infant reaches 3kg (study completion), expected within 3 months
Incidence of adverse events | 30 days post infant stopping study infant formula intake upon reaching 3kg

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Tan, Study Chair — Société des Produits Nestlé (SPN)
Locations (1):
- Tu Du Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thanh LQ, Chen Y, Hartweg M, Thi Nguyen TA. Effects of higher protein formula with improved fat blend on growth, feeding tolerance and nutritional biomarkers in preterm infants: A double-blind, randomized, controlled clinical trial. Pediatr Neonatol. 2022 May;63(3):227-238. doi: 10.1016/j.pedneo.2021.09.007. Epub 2021 Dec 4. PMID 35000893